CLINICAL TRIAL: NCT03201965
Title: A Randomized Phase 3 Study to Evaluate the Efficacy and Safety of Daratumumab in Combination With Cyclophosphamide, Bortezomib and Dexamethasone (CyBorD) Compared to CyBorD Alone in Newly Diagnosed Systemic AL Amyloidosis
Brief Title: A Study to Evaluate the Efficacy and Safety of Daratumumab in Combination With Cyclophosphamide, Bortezomib and Dexamethasone (CyBorD) Compared to CyBorD Alone in Newly Diagnosed Systemic Amyloid Light-chain (AL) Amyloidosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR108193; 54767414AMY3001 (Other: Janssen Research & Development, LLC); 2016-001737-27 (EudraCT Number); 2024-511967-26-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2017-06-27; First posted 2017-06-28 (Actual); Results first posted 2021-03-04 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Amyloidosis
MeSH Terms: conditions — Amyloidosis | interventions — Cyclophosphamide; Bortezomib; Dexamethasone; daratumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CyBorD alone (cyclophosphamide/bortezomib/dexamethasone) (Active Comparator): Participants will receive dexamethasone (40 milligrams [mg] orally or intravenous [IV] dose), followed by cyclophosphamide (300 milligram per meter square [mg/m^2] orally or IV dose), then bortezomib (1.3 mg/m^2 subcutaneous injection) weekly on Days 1, 8, 15, 22 in every 28-day cycle for a maximum of 6 cycles.
  Interventions: Drug: Cyclophosphamide; Drug: Bortezomib; Drug: Dexamethasone, 40 mg
- CyBorD plus Daratumumab (Experimental): Participants will receive dexamethasone (20 mg orally or IV dose as premedication and 20 mg on the day after daratumumab dosing) followed by 1800 mg of daratumumab subcutaneously followed by cyclophosphamide (300 mg/m^2 orally or IV dose weekly) and bortezomib (1.3 mg/m^2 subcutaneous injection weekly) on Days 1, 8, 15, 22 in every 28-day cycle for a maximum of 6 cycles. Daratumumab will be administered weekly for the first 8 weeks (2 cycles), then every 2 weeks for 4 cycles (cycles 3-6), and then every 4 weeks until progression of disease or subsequent therapy for a maximum of 2 years.
  Interventions: Drug: Daratumumab

INTERVENTIONS:
Drug: Cyclophosphamide — Participants will receive 300 mg/m^2 of cyclophosphamide as an oral or IV dose.
  Arms: CyBorD alone (cyclophosphamide/bortezomib/dexamethasone)
Drug: Bortezomib — Participants will receive 1.3 mg/m^2 of bortezomib as an subcutaneous (SC) injection.
  Arms: CyBorD alone (cyclophosphamide/bortezomib/dexamethasone)
Drug: Dexamethasone, 40 mg — Participants of CyBorD alone arm will receive 40 mg dexamethasone orally or IV dose. Participants of CyBorD plus daratumumab arm will receive dexamethasone 20 mg orally or IV dose as premedication and 20 mg on the day after daratumumab dosing to make a total of 40 mg.
  Arms: CyBorD alone (cyclophosphamide/bortezomib/dexamethasone)
Drug: Daratumumab — Participants will receive 1800 mg of daratumumab subcutaneously.
  Arms: CyBorD plus Daratumumab

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of daratumumab plus cyclophosphamide, bortezomib and dexamethasone (CyBorD) compared with CyBorD alone in treatment of newly diagnosed amyloid light chain (AL) amyloidosis participants.

DETAILED DESCRIPTION:
Participant involved in study for approx. 8 years duration includes Screening Phase (complete clinical evaluation will be done), Treatment Phase (monitoring of adverse events (AEs), laboratory abnormalities and clinical response), Post-Treatment Observation Phase (disease evaluations will be done) and a Long-term Follow-up Phase (Subsequent anticancer treatment, response to subsequent treatment, date of progression and survival status will be obtained every 16 weeks).The primary hypothesis is that daratumumab in combination with CyBorD will improve the overall complete hematological response rate compared to CyBorD alone in AL amyloidosis participants. Safety will be assessed by AEs, laboratory test results, electrocardiogram, vital sign measurements, physical examination, and Eastern Cooperative Oncology Group (ECOG) performance status.

ELIGIBILITY:
Inclusion Criteria:

* Histopathological diagnosis of amyloidosis based on detection by immunohistochemistry and polarizing light microscopy of green bi-refringent material in congo red stained tissue specimens (in an organ other than bone marrow) or characteristic electron microscopy appearance
* Measurable disease of amyloid light-chain (AL) amyloidosis as defined by at least one of the following:

  1. serum monoclonal (M)-protein greater than or equal (>=) 0.5 grams/deciliter (g/dL) by protein electrophoresis (routine serum protein electrophoresis and immunofixation [IFE] performed at a central laboratory)
  2. serum free light chain greater than or equal to (>=) 50 milligram/Liter (mg/L) with an abnormal kappa:lambda ratio or the difference between involved and uninvolved free light chains (dFLC) >= 50 mg/L
* One or more organs impacted by AL amyloidosis according to consensus guidelines
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0, 1 or 2

Exclusion Criteria:

* Prior therapy for AL amyloidosis or multiple myeloma including medications that target CD38, with the exception of 160 mg dexamethasone (or equivalent corticosteroid) maximum exposure prior to randomization
* Previous or current diagnosis of symptomatic multiple myeloma, including the presence of lytic bone disease, plasmacytomas, >= 60 percent (%) plasma cells in the bone marrow, or hypercalcemia
* Evidence of significant cardiovascular conditions as specified below:

  1. NT-ProBNP > 8500 nanogram per liter (ng/L)
  2. New York Heart Association (NYHA) classification IIIB or IV heart failure
  3. Heart failure that in the opinion of the investigator is on the basis of ischemic heart disease (eg, prior myocardial infarction with documented history of cardiac enzyme elevation and electrocardiogram [ECG] changes) or uncorrected valvular disease and not primarily due to AL amyloid cardiomyopathy
  4. Inpatient admission to a hospital for unstable angina or myocardial infarction within the last 6 months prior to first dose or percutaneous cardiac intervention with recent stent within 6 months or coronary artery bypass grafting within 6 months
  5. For participants with congestive heart failure, cardiovascular-related hospitalizations within 4 weeks prior to randomization
  6. Participants with a history of sustained ventricular tachycardia or aborted ventricular fibrillation or with a history of atrioventricular (AV) nodal or sinoatrial (SA) nodal dysfunction for which a pacemaker/implantable cardioverter-defibrillators [ICD] is indicated but not placed (participants who do have a pacemaker/ICD are allowed on study)
  7. Screening 12-lead ECG showing a baseline QT interval as corrected by Fridericia's formula (QTcF) > 500 milliseconds (msec). Participants who have a pacemaker may be included regardless of calculated QTc interval
  8. Supine systolic blood pressure < 90 millimeter of mercury (mmHg), or symptomatic orthostatic hypotension, defined as a decrease in systolic blood pressure upon standing of > 20 mmHg despite medical management (eg, midodrine, fludrocortisones) in the absence of volume depletion
* Planned stem cell transplant during the first 6 cycles of protocol therapy are excluded. Stem cell collection during the first 6 cycles of protocol therapy is permitted
* Known to be seropositive for human immunodeficiency virus (HIV)
* Any one of the following:

  1. Seropositive for hepatitis B (defined by a positive test for hepatitis B surface antigen [HBsAg]). Participants with resolved infection (ie, participants who are HBsAg negative but positive for antibodies to hepatitis B core antigen [anti-HBc] and/or antibodies to hepatitis B surface antigen [anti-HBs]) must be screened using real-time polymerase chain reaction (PCR) measurement of hepatitis B virus (HBV) deoxyribonucleic acid (DNA) levels. Those who are PCR positive will be excluded
  2. Known to be seropositive for hepatitis C (except in the setting of a sustained virologic response [SVR], defined as aviremia at least 12 weeks after completion of antiviral therapy)
* Grade 2 sensory or Grade 1 painful peripheral neuropathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 416 (Actual)
Dates: Start 2017-10-05 (Actual); Primary Completion 2020-02-14 (Actual); Study Completion 2024-11-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (139):
- United States (29):
  - Mayo Clinic Arizona, Phoenix, Arizona
  - City of Hope, Duarte, California
  - University of California San Francisco, San Francisco, California
  - Stanford University, Stanford, California
  - University of Colorado, Aurora, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Mayo Clinic, Jacksonville, Florida
  - Winship Cancer Institute Emory University, Atlanta, Georgia
  - University of Maryland, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Boston University Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Washington University School Of Medicine, St Louis, Missouri
  - Columbia University Medical Center, New York, New York
  - Weill Cornell Medical College, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - Wake Forest University Health Sciences - Cardiovascular Medicine, Winston-Salem, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - Oregon Health And Science University, Portland, Oregon
  - University of Pennsylvania Medical Center, Philadelphia, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas, MD Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Seattle Cancer Care Alliance, Seattle, Washington
- Australia (4):
  - Box Hill Hospital, Box Hill
  - Sir Charles Gairdner Hospital, Nedlands
  - Westmead Hospital, Westmead
  - Princess Alexandra Hospital, Woolloongabba
- Belgium (4):
  - Institut Jules Bordet, Anderlecht
  - UZ Gent, Ghent
  - Az Groeninge, Kortrijk
  - Universitair Ziekenhuis Leuven, Leuven
- Brazil (8):
  - Hospital das Clinicas de Porto Alegre, Porto Alegre
  - Sociedade Pernambucana de Combate ao Cancer, Recife
  - Instituto de Educacao, Pesquisa e Gestao em Saude Instituto Americas (COI), Rio de Janeiro
  - Hospital Sao Rafael, Salvador
  - Fundacao Faculdade Regional de Medicina de Sao Jose do Rio Preto Hospital de Base, São José do Rio Preto
  - Clinica Sao Germano, São Paulo
  - Instituto de Assistencia Medica ao Servidor Publico Estadual IAMSPE, São Paulo
  - Hospital Das Clinicas Da Faculdade De Medicina Da USP, São Paulo
- Canada (6):
  - Arthur J E Child Comprehensive Cancer Centre, Calgary, Alberta
  - Alberta Health Services, Edmonton, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - London Health Sciences Center, London, Ontario
  - University Health Network UHN Princess Margaret Cancer Centre, Toronto, Ontario
  - McGill University Health Centre, Montreal, Quebec
- China (5):
  - Peking University First Hospital, Beijing
  - Peking University People s Hospital, Beijing
  - First affiliated Hospital of Zhejiang University, Hangzhou
  - Ruijin Hospital Shanghai Jiao Tong University, Shanghai
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou
- Denmark (3):
  - Aarhus University Hospital, Aarhus N
  - Dep. of Hematology, Rigshospitalet, Copenhagen
  - Odense Universitets Hospital, Odense
- France (11):
  - CHU Dijon, Dijon
  - Hopital Claude Huriez, Lille
  - CHU de Limoges - Fédération Hépatologie, Limoges
  - Institut Paoli Calmettes, Marseille
  - Chu Hotel Dieu, Nantes
  - Hopital Saint Louis, Paris
  - Centre hospitalier Lyon-Sud, Pierre-Bénite
  - CHU De Poitiers, Poitiers
  - CHU Rangueil, Toulouse
  - CHU Bretonneau, Tours
  - CHU de Nancy_ Hopital Brabois, Vandœuvre-lès-Nancy
- Germany (7):
  - Charite Campus Benjamin Franklin, Berlin
  - Heinrich-Heine-Universität Düsseldorf, Düsseldorf
  - Universitatsklinikum Essen, Essen
  - HOPA-Hämatologisch-Onkologische Praxis Altona MVZ GmbH, Hamburg
  - Universitaetsklinikum Heidelberg Medizinische Klinik V, Heidelberg
  - Universitaetsklinikum Tuebingen der Eberhard-Karls-Universitaet, Abteilung fuer Innere Medizin II,, Tübingen
  - Universitätsklinikum Würzburg Med. Klinik U. Poliklinik Ii, Würzburg
- Greece (2):
  - Alexandra General Hospital of Athens, Athens
  - University General Hospital of Rio, Pátrai
- Hungary (2):
  - Semmelweis Egyetem I.Belgyogyaszati Klinika, Budapest
  - Del Pesti Centrumkorhaz Orszagos Hematologiai es Infektologiai Intezet Szent Laszlo Telephely, Budapest
- Israel (5):
  - Carmel Hospital, Haifa
  - Hadassah Medical Center, Jerusalem
  - Sheba Medical Center, Ramat Gan
  - Sourasky Medical Center, Tel Aviv
  - Assaf Ha'Rofeh Medical Center, Ẕerifin
- Italy (6):
  - Policlinico di Bari, Bari
  - Istituto di Ematologia Seràgnoli azienda ospedaliera univeristaria Policlinico S.Orsola-Malpighi, Bologna
  - Casa di Cura La Maddalena, Palermo
  - Amyloidosis Research and Treatment Center, Fondazione IRCCS Policlinico San Matteo, Pavia
  - Dipartimento Di Biotecnologie Cellulari Ed Ematologia-Università ''La Sapienza'',Policlinico Umberto I, Roma
  - A.O.U. Città della Salute e della Scienza, Torino
- Japan (12):
  - Fukushima Medical University Hospital, Fukushima
  - Hiroshima Red Cross Hospital & Atomic-bomb Survivors Hospital, Hiroshima
  - Teine Keijinkai Hospital, Hokkaido
  - Kanazawa University Hospital, Kanazawa
  - Kumamoto University Hospital, Kumamoto
  - Kyoto Kuramaguchi Medical Center, Kyoto
  - Shinshu University Hospital, Matsumoto
  - Matsuyama Red Cross Hospital, Matsuyama
  - Nagoya City University Hospital, Nagoya
  - National Hospital Organization Okayama Medical Center, Okayama
  - Japanese Red Cross Medical Center, Shibuya City
  - Tokushima University Hospital, Tokushima
- Mexico (2):
  - Centro de Investigación Farmacéutica Especializada, Guadalajara
  - Hospital Universitario Dr Jose Eleuterio Gonzalez, Monterrey
- Netherlands (5):
  - UMCG, Groningen
  - Erasmus MC, Rotterdam
  - Haga ziekenhuis, The Hague
  - UMC Utrecht, Utrecht
  - Maxima Medisch Centrum, Veldhoven
- Poland (3):
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej Zespol Szpitali Miejskich, Chorzów
  - SKPP UM w Poznaniu, Poznan
  - Instytut Hematologii i Transfuzjologii, Warsaw
- South Korea (5):
  - Pusan National University Hospital, Busan
  - Seoul National University Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea Seoul St Marys Hospital, Seoul
- Spain (10):
  - Inst. Cat. D'Oncologia-Badalona, Badalona
  - Hosp Univ Vall D Hebron, Barcelona
  - Hosp Clinic de Barcelona, Barcelona
  - Hosp. Univ. Ramon Y Cajal, Madrid
  - Hosp Univ Fund Jimenez Diaz, Madrid
  - Hosp. Univ. 12 de Octubre, Madrid
  - Clinica Univ. de Navarra, Pamplona
  - Hosp Clinico Univ de Salamanca, Salamanca
  - Hosp. Univ. de Canarias, San Cristóbal de La Laguna
  - Hosp. Univ. Dr. Peset, Valencia
- Sweden (2):
  - South Elvsborg Hospital, Borås
  - Skanes universitetssjukhus, Lund
- Turkey (Türkiye) (6):
  - Ankara Universitesi Tip Fakultesi Cebeci Hastanesi, Ankara
  - Akdeniz University Medical Faculty, Antalya
  - Ondokuz Mayis Universitesi Tip Fakultesiy, Atakum
  - Istanbul University Istanbul Medical Faculty, Istanbul
  - Dokuz Eylul Universitesi Tip Fakultesi, Izmir
  - Erciyes University Medical Faculty, Talas
- United Kingdom (2):
  - University Hospitals Birmingham NHS Trust,, Birmingham
  - University College Hospital, London

REFERENCES:
- [Derived] Suzuki K, Wechalekar AD, Kim K, Shimazaki C, Kim JS, Ikezoe T, Min CK, Zhou F, Cai Z, Chen X, Iida S, Katoh N, Fujisaki T, Shin HJ, Tran N, Qin X, Vasey SY, Tromp B, Weiss BM, Comenzo RL, Kastritis E, Lu J. Daratumumab plus bortezomib, cyclophosphamide, and dexamethasone in Asian patients with newly diagnosed AL amyloidosis: subgroup analysis of ANDROMEDA. Ann Hematol. 2023 Apr;102(4):863-876. doi: 10.1007/s00277-023-05090-z. Epub 2023 Mar 2. PMID 36862168
- [Derived] Minnema MC, Dispenzieri A, Merlini G, Comenzo RL, Kastritis E, Wechalekar AD, Grogan M, Witteles R, Ruberg FL, Maurer MS, Tran N, Qin X, Vasey SY, Weiss BM, Vermeulen J, Jaccard A. Outcomes by Cardiac Stage in Patients With Newly Diagnosed AL Amyloidosis: Phase 3 ANDROMEDA Trial. JACC CardioOncol. 2022 Nov 15;4(4):474-487. doi: 10.1016/j.jaccao.2022.08.011. eCollection 2022 Nov. PMID 36444227
- [Derived] Kastritis E, Palladini G, Minnema MC, Wechalekar AD, Jaccard A, Lee HC, Sanchorawala V, Gibbs S, Mollee P, Venner CP, Lu J, Schonland S, Gatt ME, Suzuki K, Kim K, Cibeira MT, Beksac M, Libby E, Valent J, Hungria V, Wong SW, Rosenzweig M, Bumma N, Huart A, Dimopoulos MA, Bhutani D, Waxman AJ, Goodman SA, Zonder JA, Lam S, Song K, Hansen T, Manier S, Roeloffzen W, Jamroziak K, Kwok F, Shimazaki C, Kim JS, Crusoe E, Ahmadi T, Tran N, Qin X, Vasey SY, Tromp B, Schecter JM, Weiss BM, Zhuang SH, Vermeulen J, Merlini G, Comenzo RL; ANDROMEDA Trial Investigators. Daratumumab-Based Treatment for Immunoglobulin Light-Chain Amyloidosis. N Engl J Med. 2021 Jul 1;385(1):46-58. doi: 10.1056/NEJMoa2028631. PMID 34192431
- [Derived] Palladini G, Kastritis E, Maurer MS, Zonder J, Minnema MC, Wechalekar AD, Jaccard A, Lee HC, Bumma N, Kaufman JL, Medvedova E, Kovacsovics T, Rosenzweig M, Sanchorawala V, Qin X, Vasey SY, Weiss BM, Vermeulen J, Merlini G, Comenzo RL. Daratumumab plus CyBorD for patients with newly diagnosed AL amyloidosis: safety run-in results of ANDROMEDA. Blood. 2020 Jul 2;136(1):71-80. doi: 10.1182/blood.2019004460. PMID 32244252

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants with newly diagnosed Amyloid Light-chain (AL) amyloidosis with measurable disease and at least one organ involvement, and Mayo cardiac stage I - IIIA, who had not received prior therapy for AL amyloidosis or multiple myeloma were enrolled.
Groups:
- Run-In: Daratumumab Plus CyBorD: Participants received the combination therapy during Run-in phase starting with 20 milligrams (mg) dexamethasone as premedication followed by daratumumab 1800 mg on Day 1 Cycle 1, then cyclophosphamide 300 milligram per meter square (mg/m^2) orally or intravenous (IV) maximum weekly dose 500 mg, followed by bortezomib 1.3 mg/m^2 subcutaneous (SC) injection once every week and dexamethasone remaining 20 mg post daratumumab dosing for up to 1 cycle (28 Days) to assess the safety before randomizing participants in CyBorD or daratumumab plus CyBorD arms. However, participants also continued daratumumab plus CyBorD for up to 6 cycles and then daratumumab monotherapy for up to 24 months from the start of treatment. After completion of treatment phase participants entered into the post treatment observation phase and were continued with disease evaluations every 8 weeks post last dose up to disease progression (up to 6.5 years). Participants then entered into long term follow up phase and were followed up for survival every 16 weeks (up to 7.1 years).
- CyBorD: Participants received dexamethasone (40 mg weekly dose)starting from cycle 1 day1 in every 28-day cycle followed by cyclophosphamide 300 mg/m^2 orally or IV maximum weekly dose 500 mg and then bortezomib 1.3 mg/m^2 SC injection once weekly up to 7.33 months. All cycles were of 28 days. After completion of treatment phase participants entered into the post treatment observation phase and were continued with disease evaluations every 8 weeks post last dose up to disease progression (up to 6.5 years). Participants then entered into long term follow up phase and were followed up for survival every 16 weeks (up to 7.1 years).
- Daratumumab Plus CyBorD: Participants received combination therapy for six cycles of 28 days each, daratumumab 1800 mg SC weekly starting from cycles 1 day 1 and cycle 2, every 2 weeks in cycles 3 through 6, dexamethasone 40 mg weekly (on days of daratumumab dosing, dexamethasone was split, 20 mg as premedication and 20 mg as post daratumumab dosing), cyclophosphamide 300 mg/m^2 orally or IV maximum weekly dose 500 mg, bortezomib 1.3 mg/m^2 SC injection once weekly. After 6 cycles, participants continued to receive daratumumab SC monotherapy until disease progression, start of subsequent therapy or up to 26.71 months from the first dose of study treatment. All cycles were of 28 days. After completion of treatment phase participants entered into the post treatment observation phase and were continued with disease evaluations every 8 weeks post last dose up to disease progression (up to 6.5 years). Participants then entered into long term follow up phase and were followed up for survival every 16 weeks (up to 7.1 years).
Period: Overall Study
Arm/Group | Run-In: Daratumumab Plus CyBorD | CyBorD | Daratumumab Plus CyBorD
Started | 28 | 193 | 195
Treated | 28 | 188 | 193
Completed | 0 | 0 | 0
Not Completed | 28 | 193 | 195
Not completed — Death | 5 | 65 | 47
Not completed — Lost to Follow-up | 0 | 6 | 0
Not completed — Withdrawal by Subject | 3 | 23 | 8
Not completed — Sponsor's Decision | 20 | 99 | 140

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Run-In: Daratumumab Plus CyBorD | CyBorD | Daratumumab Plus CyBorD | Total
Number analyzed (Participants) | 28 | 193 | 195 | 416
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.8 (11.2) | 64 (9.66) | 62.2 (10.16) | 63.2 (10.03)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 11 | 76 | 87 | 174
  Male | 16 | 117 | 108 | 241
  Undifferentiated Sex | 1 | 0 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 13 | 9 | 23
  Not Hispanic or Latino | 26 | 176 | 179 | 381
  Unknown or Not Reported | 1 | 4 | 7 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 1 | 3
  Asian | 0 | 34 | 30 | 64
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 2 | 7 | 6 | 15
  White | 25 | 143 | 151 | 319
  More than one race | 0 | 1 | 0 | 1
  Unknown or Not Reported | 1 | 5 | 7 | 13
Region of Enrollment [Count of Participants; unit: Participants]
  AUSTRALIA | 0 | 15 | 12 | 27
  BELGIUM | 0 | 1 | 2 | 3
  BRAZIL | 0 | 7 | 4 | 11
  CANADA | 0 | 10 | 9 | 19
  CHINA | 0 | 6 | 6 | 12
  DENMARK | 0 | 1 | 1 | 2
  FRANCE | 0 | 22 | 16 | 38
  GERMANY | 0 | 11 | 8 | 19
  GREECE | 0 | 11 | 16 | 27
  HUNGARY | 0 | 2 | 2 | 4
  ISRAEL | 0 | 5 | 6 | 11
  ITALY | 0 | 5 | 4 | 9
  JAPAN | 0 | 13 | 15 | 28
  MEXICO | 0 | 1 | 1 | 2
  NETHERLANDS | 0 | 4 | 7 | 11
  POLAND | 0 | 2 | 2 | 4
  SOUTH KOREA | 0 | 12 | 8 | 20
  SPAIN | 0 | 11 | 21 | 32
  SWEDEN | 0 | 2 | 1 | 3
  TURKEY | 0 | 7 | 10 | 17
  UNITED KINGDOM | 0 | 4 | 4 | 8
  UNITED STATES | 28 | 41 | 40 | 109
Weight group in Kilograms (Kg) [Count of Participants; unit: Participants]
  <=65 kg | 5 | 74 | 62 | 141
  >65 to 85 kg | 12 | 74 | 96 | 182
  >85 kg | 11 | 45 | 37 | 93
Baseline Major Organ Involvement [Count of Participants; unit: Participants] — Organ involvement assessment: biopsy. Heart: echo: mean wall thickness greater than (>) 12 millimeter, no other cardiac cause; kidney: 24- hour urine protein >0.5 gram per day, predominantly albumin; liver: total liver span >15 centimeter in absence of heart failure or alkaline phosphatase >1.5 times institutional upper limit of normal.
  Participants
    Baseline Organ Involvement: Heart | 17 | 137 | 140 | 294
    Baseline Organ Involvement: Kidney | 19 | 114 | 115 | 248
    Baseline Organ Involvement: Liver | 4 | 16 | 15 | 35
Number of Organs Involved [Mean (Standard Deviation); unit: organs] | 2.0 (0.881) | 2.0 (1.03) | 2.0 (0.97) | 2.0 (0.99)
Number of Organs Involved [Count of Participants; unit: Participants] — Number of participants whose 1 organ, 2 organs, 3 or more than 3 organs involved at baseline was reported. Organs like heart, kidney, and liver were considered.
  Participants
    1 Organ | 9 | 68 | 66 | 143
    2 Organs | 13 | 77 | 76 | 166
    >=3 Organ | 6 | 48 | 53 | 107
Cardiac Stage Based on Mayo Clinic Cardiac Staging System [Count of Participants; unit: Participants] — Cardiac stage is derived based on the combination of NT-proBNP (N-terminal pro b-type natriuretic peptide) and hs-cTnT (high sensitivity cardiac troponin T). Risk factor includes NT-proBNP >332 nanogram per liter (ng/L) and Hs-cTnT >54 ng/L. Stage I includes no markers above the cutoff, stage 2 includes one marker above the cutoff, stage 3a includes both markers above the cutoff, and stage 3b includes NT-proBNP >8500 ng/L and hs-cTnT >54 ng/L.
  Participants
    Class I | 6 | 43 | 47 | 96
    Class II | 16 | 80 | 76 | 172
    Class IIIa | 5 | 64 | 70 | 139
    Class IIIb | 1 | 6 | 2 | 9
New York Heart Association (NYHA) Class [Count of Participants; unit: Participants] — The NYHA classification: Class I- No symptoms and no limitation in ordinary physical activity, example, shortness of breath when walking, climbing stairs; class II- mild symptoms (mild shortness of breath and/or angina) and slight limitation during ordinary activity; class IIIA- marked limitation in activity due to symptoms, even during less than ordinary activity, example, walking short distances (20-100 meter).Comfortable only at rest.
  Participants
    Class I | 17 | 94 | 101 | 212
    Class II | 10 | 89 | 77 | 176
    Class IIIA | 1 | 10 | 17 | 28

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Overall Complete Hematologic Response (CHR)
Description: Overall CHR rate was defined as percentage of participants who achieved CHR, according to the International Amyloidosis Consensus Criteria. CHR: normalization of free light chain levels and ratio, negative serum, and urine immunofixation. If involved free light chain (iFLC) is less than (<) upper limit of normal (ULN) and serum and urine Immunofixation electrophoresis (IFE) are negative, then neither a normal uninvolved free light chain (uFLC) level nor a normal free light chain (FLC) ratio are required for complete response (CR).
Time Frame: Up to 2.4 years
Population: The intent to treat analysis set included all the participants who were randomized and received at least one dose of study treatment in the study. Data for this outcome measure (OM) was planned to be collected and analyzed for specified arms only.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CyBorD | Daratumumab Plus CyBorD
Number analyzed (Participants) | 193 | 195
percentage of participants | 18.1 [13.0 to 24.3] | 53.3 [46.1 to 60.5]
Statistical Analysis 1: Comparison: CyBorD vs Daratumumab Plus CyBorD; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 5.13, 95% CI 2-sided [3.22 to 8.16]

2. Secondary Outcome: Major Organ Deterioration Progression-Free Survival (MOD-PFS)
Description: MOD-PFS was defined as duration from the date of randomization to either hematologic progression, or major organ deterioration (clinical manifestation of cardiac failure or renal failure), or death, whichever occurred first. Per international amyloidosis consensus criteria (IACC), hematologic progression was defined as satisfying any one of the following criteria: 1) From CHR, abnormal free light chain ratio (light chain must be double and >ULN); 2) From CHR/VGPR/PR, 50 percent (%) increase in serum M-protein to >0.5 grams per deciliter (g/dL) or 50% increase in urine M-protein to 200 milligrams (mg)/day; 3) free light chain increase of 50% to 100 milligrams (mg)/Liter (L).
Time Frame: From date of first randomization (Day -3) upto 6.5 years
Population: The intent to treat analysis set included all randomized participants. Data for this outcome measure was planned to be collected and analyzed for specified arms only.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | CyBorD | Daratumumab Plus CyBorD
Number analyzed (Participants) | 193 | 195
months | 30.23 [16.66 to 48.89] | NA [NA to NA] — Here, 'NA' signifies that Median, lower limit and upper limit of 95% confidence interval (CI) could not be estimated due to an insufficient number of participants with events.

3. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) was measured from the date of randomization to the date of the participant's death.
Time Frame: From date of first randomization (Day -3) up to 7.1 years
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | CyBorD | Daratumumab Plus CyBorD
Number analyzed (Participants) | 193 | 195
Months | NA [NA to NA] — Here, 'NA' signifies that median, lower limit and upper limit of 95% CI could not be estimated due to an insufficient number of participants with events. | NA [NA to NA] — Here, 'NA' signifies that median, lower limit and upper limit of 95% CI could not be estimated due to an insufficient number of participants with events.

4. Secondary Outcome: Organ Response Rate (OrRR) at 6 Months: Cardiac Response
Description: The Organ Response Rate (OrRR) for heart was defined as the percentage of participants with baseline involvement of the heart who achieved a confirmed organ response in the heart. Cardiac response was defined as as a decrease of >30% in N-terminal pro-B-type natriuretic peptide (NT-proBNP) levels and greater than (>)300 nanogram/Litre (ng/L).
Time Frame: Month 6
Population: Cardiac response-evaluable participants had baseline NT-proBNP >=650 ng/L or NYHA class 3 or 4, plus received at least 1 administration of study treatment and had at least one post-baseline. NT-proBNP measurement (if baseline NT-proBNP >=650 nanograms per liter [ng/L]) or NYHA function evaluation (if baseline NYHA class 3 or 4). Data for this outcome measure was planned to be collected and analyzed for specified arms only.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | CyBorD | Daratumumab Plus CyBorD
Number analyzed (Participants) | 117 | 118
Percentage of participants | 22.2 [15.1 to 30.8] | 41.5 [32.5 to 51.0]

5. Secondary Outcome: Organ Response Rate (OrRR) at 6 Months: Renal Response
Description: The OrRR for kidney was defined as the percentage of participants with baseline involvement of the kidney who achieved a confirmed renal response in the kidney. Renal response was defined as more than equal to (≥) 30% decrease in proteinuria or proteinuria decreased to <0.5 grams (g)/24 hours in the absence of renal progression.
Time Frame: Month 6
Population: Renal response-evaluable participants had baseline urine protein >0.5 g/day, received at least one administration of study treatment, and had at least post-baseline urine protein measurement. Data for this outcome measure was planned to be collected and analyzed for specified arms only.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | CyBorD | Daratumumab Plus CyBorD
Number analyzed (Participants) | 113 | 117
Percentage of participants | 27.4 [19.5 to 36.6] | 53.8 [44.4 to 63.1]

6. Secondary Outcome: Organ Response Rate (OrRR) at 6 Months: Liver Response
Description: The OrRR for liver was defined as the percentage of participants with baseline involvement of the liver who achieved a confirmed liver response in the liver. Liver response was defined as 50% decrease in abnormal alkaline phosphatase value.
Time Frame: Month 6
Population: Liver response-evaluable participants had baseline abnormal alkaline phosphatase >1.5*upper limit of normal (ULN), at least 1 administration of study treatment and had at least one post-baseline alkaline phosphatase measurement. Data for this outcome measure was planned to be collected and analyzed for specified arms.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | CyBorD | Daratumumab Plus CyBorD
Number analyzed (Participants) | 14 | 10
Percentage of participants | 7.1 [0.2 to 33.9] | 40.0 [12.2 to 73.8]

7. Secondary Outcome: Percentage of Participants Who Achieved Complete Hematologic Response (CHR) at 6 Months
Description: CHR rate was defined as percentage of participants who achieved CHR, according to the International Amyloidosis Consensus Criteria. CHR: normalization of free light chain levels and ratio, negative serum, and urine immunofixation. If involved free light chain is < ULN and serum and urine IFE are negative, then neither a normal uninvolved free light chain (uFLC) level nor a normal free light chain (FLC) ratio are required for Complete Response (CR).
Time Frame: Month 6
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | CyBorD | Daratumumab Plus CyBorD
Number analyzed (Participants) | 193 | 195
Percentage of participants | 14.0 [9.4 to 19.7] | 50.3 [43.0 to 57.5]

8. Secondary Outcome: Time to Complete Hematologic Response (CHR)
Description: Time to CHR was defined as time between the date of randomization and first efficacy evaluation at which the participant has met all criteria for hematologic CR. CHR was primarily defined by negative immunofixation results and normalized free light chain (FLC) parameters.
Time Frame: From date of first randomization (Day -3) up to 6.5 years
Population: Responders in intent to-treat analysis set included participants of intent to-treat analysis set who had hematologic response (complete hematologic response, VGPR and PR). Here, 'N' (number of participants analyzed) signifies number of participants evaluable for this outcome measure. Data for this outcome measure was planned to be collected and analyzed for specified arms only.
Measure: Median (Full Range); unit: Days
Arm/Group | CyBorD | Daratumumab Plus CyBorD
Number analyzed (Participants) | 37 | 116
Days | 85.00 [14.0 to 617.0] | 67.50 [8.0 to 879.0]

9. Secondary Outcome: Time to Cardiac Response
Description: Time to cardiac response was defined as the time between the date of randomization and the first efficacy evaluation at which the participant had cardiac response.
Time Frame: From date of first randomization (Day -3) up to 6.5 years
Population: Cardiac response-evaluable participants had baseline NT-proBNP greater than equal to >= 650 ng/L or NYHA class 3/4, with at least one post-baseline NT-proBNP or NYHA assessment after receiving treatment. Here, 'N' (number of participants analyzed) signifies number of participants evaluable for this outcome measure. Data for this outcome measure was planned to be collected and analyzed for specified arms.
Measure: Median (Full Range); unit: Months
Arm/Group | CyBorD | Daratumumab Plus CyBorD
Number analyzed (Participants) | 49 | 75
Months | 4.67 [0.9 to 25.5] | 3.84 [1.0 to 17.8]

10. Secondary Outcome: Time to Liver Response
Description: Time to liver response was defined as the time between the date of randomization and the first efficacy evaluation at which the participant had liver response.
Time Frame: From date of first randomization (Day -3) up to 6.5 years
Population: Liver response-evaluable participant had alkaline phosphatase >1.5*ULN, received treatment, and had a post-baseline test. Here, 'N' (number of participants analyzed) signifies number of participants evaluable for this outcome measure. Data for this outcome measure was planned to be collected and analyzed for specified arms only.
Measure: Median (Full Range); unit: Months
Arm/Group | CyBorD | Daratumumab Plus CyBorD
Number analyzed (Participants) | 3 | 6
Months | 10.61 [2.0 to 15.2] | 4.68 [1.0 to 22.6]

11. Secondary Outcome: Time to Renal Response
Description: Time to renal response was defined as the time between the date of randomization and the first efficacy evaluation at which the participant had renal response.
Time Frame: From date of first randomization (Day -3) up to 6.5 years
Population: Renal response-evaluable participants had urine protein >0.5 g/day at baseline, received treatment, and had a postbaseline urine test. Here, 'N' (number of participants analyzed) signifies number of participants evaluable for this outcome measure. Data for this outcome measure was planned to be collected and analyzed for specified arms only.
Measure: Median (Full Range); unit: Months
Arm/Group | CyBorD | Daratumumab Plus CyBorD
Number analyzed (Participants) | 55 | 96
Months | 3.75 [0.9 to 42.2] | 1.91 [0.4 to 38.3]

12. Secondary Outcome: Time to Subsequent Non-cross Resistant Anti-plasma Cell Therapy
Description: Time to subsequent non-cross resistant anti-plasma cell therapy was defined as the time from the date of randomization to the start date of subsequent non-cross resistant, anti-plasma cell therapy.
Time Frame: From date of first randomization (Day -3) up to 6.5 years
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | CyBorD | Daratumumab Plus CyBorD
Number analyzed (Participants) | 193 | 195
Months | 11.30 [8.71 to 21.03] | NA [NA to NA] — Here, 'NA' signifies that median, lower limit and upper limit of 95% CI could not be estimated due to an insufficient number of participants with events.

13. Secondary Outcome: Duration of Complete Hematologic Response (CHR)
Description: Duration of CHR was defined as the time between the date of initial documentation of CHR to the date of first documented evidence of hematologic progressive diseased. CHR was primarily defined by negative immunofixation results and normalized FLC parameters.
Time Frame: From date of first randomization (Day -3) up to 6.5 years
Population: Responders in intent-to-treat analysis set included all randomized participants. Here, 'N' (number of participants analyzed) signifies number of participants evaluable for this outcome measure. Data for this outcome measure was planned to be collected and analyzed for specified arms only.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | CyBorD | Daratumumab Plus CyBorD
Number analyzed (Participants) | 37 | 116
Months | NA [56.74 to NA] — Here, 'NA' signifies that Median and upper limit of 95% CI could not be estimated due to an insufficient number of participants with events. | NA [NA to NA] — Here, 'NA' signifies that Median, lower limit and upper limit of 95% CIcould not be estimated due to an insufficient number of participants with events.

14. Secondary Outcome: Hematologic Very Good Partial Response (VGPR) or Better Rate
Description: Hematologic VGPR or Better Rate was defined as percentage of participants who achieved hematologic Complete response (CR) or VGPR. VGPR was defined as the difference between involved iFLC and uFLC after treatment for baseline difference between iFLC and uFLC (dFLC) >50 milligrams per liter (mg/L): Reduction in the dFLC <40 mg/L. For Baseline dFLC < 50 mg/L: more than (>) 90% reduction in serum M-protein plus urine M-protein <100 mg/24 hours. CR was negative immunofixation on the serum and urine, and disappearance of any soft tissue plasmacytomas, and < 5% PCs in bone marrow.
Time Frame: From date of first randomization (Day -3) up to 6.5 years
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | CyBorD | Daratumumab Plus CyBorD
Number analyzed (Participants) | 193 | 195
Percentage of participants | 50.3 [43.0 to 57.5] | 79.0 [72.6 to 84.5]

15. Secondary Outcome: Change From Baseline in the European Organisation for Research and Treatment of Cancer - Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) Fatigue
Description: The EORTC-QLQ-C30 a 30-question tool was used to assess the overall quality of life (QoL) in cancer patients. It included 30 items resulting in 5 functional scales (physical, role, emotional, cognitive, and social functioning), 1 Global health status (GHS) scale, 3 symptom scales (fatigue, nausea and vomiting, and pain), and 6 single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). The questionnaire includes 28 items with 4-point Likert type responses from "1-not at all" to "4-very much" to assess functioning and symptoms; 2 items with 7-point Likert scales (1= poor and 7= excellent) for global health and overall QoL. Scores were transformed to a 0 to 100 scale, with higher scores representing better GHS, better functioning, and more symptoms.
Time Frame: Baseline (Day -28), Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 76, 80, 84, 88, 92 and 96
Population: The intent to treat analysis set included all randomized participants. Here 'N' (number of participants analyzed) signifies number of participants who were evaluable for this outcome measure. Here 'n' (number analyzed) signifies number of participants analyzed at specified timepoints. Data for this outcome measure was planned to be collected and analyzed for specified arms only.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on scale
Arm/Group | CyBorD | Daratumumab Plus CyBorD
Number analyzed (Participants) | 178 | 179
Score on scale
  Week 4: number analyzed (Participants) | 155 | 155
  Week 4 | 3.79 [0.33 to 7.25] | 2.07 [-1.39 to 5.53]
  Week 8: number analyzed (Participants) | 146 | 152
  Week 8 | 4.04 [0.50 to 7.58] | 3.93 [0.44 to 7.42]
  Week 12: number analyzed (Participants) | 137 | 137
  Week 12 | 6.35 [2.74 to 9.96] | 2.77 [-0.82 to 6.37]
  Week 16: number analyzed (Participants) | 130 | 132
  Week 16 | 9.92 [6.25 to 13.60] | 1.54 [-2.10 to 5.17]
  Week 20: number analyzed (Participants) | 114 | 137
  Week 20 | 6.83 [3.01 to 10.65] | 3.87 [0.27 to 7.47]
  Week 24: number analyzed (Participants) | 33 | 127
  Week 24 | 0.69 [-5.40 to 6.79] | 0.30 [-3.37 to 3.98]
  Week 28: number analyzed (Participants) | 85 | 27
  Week 28 | 3.30 [-0.90 to 7.51] | 2.14 [-4.41 to 8.69]
  Week 32: number analyzed (Participants) | 15 | 105
  Week 32 | -3.14 [-11.77 to 5.49] | -4.92 [-8.82 to -1.03]
  Week 36: number analyzed (Participants) | 8 | 20
  Week 36 | -10.25 [-21.95 to 1.45] | -12.59 [-20.06 to -5.13]
  Week 40: number analyzed (Participants) | 12 | 100
  Week 40 | 2.09 [-7.49 to 11.68] | -5.39 [-9.34 to -1.43]
  Week 44: number analyzed (Participants) | 9 | 19
  Week 44 | 1.57 [-9.46 to 12.59] | -9.55 [-17.19 to -1.90]
  Week 48: number analyzed (Participants) | 32 | 94
  Week 48 | -2.82 [-8.98 to 3.34] | -7.99 [-12.03 to -3.95]
  Week 52: number analyzed (Participants) | 20 | 23
  Week 52 | -1.69 [-9.28 to 5.90] | -5.56 [-12.58 to 1.46]
  Week 56: number analyzed (Participants) | 178 | 88
  Week 56 | -1.88 [-10.00 to 6.24] | -6.77 [-10.89 to -2.64]
  Week 60: number analyzed (Participants) | 16 | 24
  Week 60 | -2.62 [-10.99 to 5.75] | -9.23 [-16.12 to -2.34]
  Week 64: number analyzed (Participants) | 12 | 81
  Week 64 | -3.55 [-13.13 to 6.04] | -10.36 [-14.61 to -6.12]
  Week 68: number analyzed (Participants) | 10 | 34
  Week 68 | 0.84 [-9.63 to 11.30] | -5.96 [-11.90 to -0.03]
  Week 72: number analyzed (Participants) | 23 | 75
  Week 72 | -0.44 [-7.55 to 6.67] | -11.80 [-16.16 to -7.45]
  Week 76: number analyzed (Participants) | 12 | 31
  Week 76 | -5.08 [-14.68 to 4.51] | -8.91 [-15.07 to -2.75]
  Week 80: number analyzed (Participants) | 24 | 79
  Week 80 | -6.00 [-12.96 to 0.97] | -10.79 [-15.07 to -6.51]
  Week 84: number analyzed (Participants) | 8 | 30
  Week 84 | -17.23 [-28.87 to -5.58] | -10.39 [-16.63 to -4.14]
  Week 88: number analyzed (Participants) | 12 | 80
  Week 88 | -6.71 [-16.34 to 2.91] | -9.83 [-14.08 to -5.57]
  Week 92: number analyzed (Participants) | 7 | 29
  Week 92 | -7.43 [-19.78 to 4.92] | -12.11 [-18.43 to -5.78]
  Week 96: number analyzed (Participants) | 178 | 64
  Week 96 | -5.75 [-13.87 to 2.37] | -8.56 [-13.16 to -3.95]

16. Secondary Outcome: Change From Baseline in the Short Form Health Survey, Version 2, the Mental Component Summary, (SF-36v2 MCS)
Description: The SF-36 Health Survey was a generic measure of health status. The SF-36 consisted of 36 questions that yield an eight-scale (physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health) profile of functional health and well-being, as well as 2 physical and mental health summary measures and a preference-based health utility index. The physical component summary (PCS), the mental component summary (MCS), and the 8 domain scores range from zero (0) to 100, with higher scores representing higher level of functioning.
Time Frame: as for outcome 15
Population: as for outcome 15
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on scale
Arm/Group | CyBorD | Daratumumab Plus CyBorD
Number analyzed (Participants) | 176 | 176
Score on scale
  Week 4: number analyzed (Participants) | 150 | 148
  Week 4 | -0.43 [-1.95 to 1.09] | -0.19 [-1.71 to 1.34]
  Week 8: number analyzed (Participants) | 143 | 144
  Week 8 | -1.09 [-2.64 to 0.46] | -1.42 [-2.96 to 0.12]
  Week 12: number analyzed (Participants) | 135 | 135
  Week 12 | -1.86 [-3.44 to -0.28] | -0.17 [-1.74 to 1.40]
  Week 16: number analyzed (Participants) | 128 | 130
  Week 16 | -3.15 [-4.76 to -1.54] | -0.35 [-1.94 to 1.23]
  Week 20: number analyzed (Participants) | 111 | 134
  Week 20 | -2.36 [-4.04 to -0.68] | -0.42 [-1.99 to 1.16]
  Week 24: number analyzed (Participants) | 32 | 125
  Week 24 | -1.84 [-4.50 to 0.82] | -0.60 [-2.20 to 1.01]
  Week 28: number analyzed (Participants) | 83 | 27
  Week 28 | -3.26 [-5.10 to -1.42] | -0.93 [-3.74 to 1.88]
  Week 32: number analyzed (Participants) | 15 | 103
  Week 32 | 0.19 [-3.51 to 3.89] | 0.61 [-1.09 to 2.31]
  Week 36: number analyzed (Participants) | 8 | 19
  Week 36 | -0.45 [-5.47 to 4.57] | 1.22 [-2.05 to 4.49]
  Week 40: number analyzed (Participants) | 12 | 99
  Week 40 | -0.56 [-4.67 to 3.54] | 2.02 [0.30 to 3.74]
  Week 44: number analyzed (Participants) | 8 | 19
  Week 44 | 1.30 [-3.70 to 6.30] | 1.55 [-1.73 to 4.82]
  Week 48: number analyzed (Participants) | 32 | 92
  Week 48 | 0.26 [-2.39 to 2.91] | 2.18 [0.41 to 3.94]
  Week 52: number analyzed (Participants) | 20 | 22
  Week 52 | 0.69 [-2.57 to 3.94] | 1.33 [-1.73 to 4.39]
  Week 56: number analyzed (Participants) | 176 | 87
  Week 56 | -0.35 [-3.83 to 3.13] | 0.91 [-0.88 to 2.71]
  Week 60: number analyzed (Participants) | 16 | 24
  Week 60 | 2.20 [-1.39 to 5.79] | 1.32 [-1.64 to 4.28]
  Week 64: number analyzed (Participants) | 11 | 80
  Week 64 | -2.00 [-6.28 to 2.28] | 2.74 [0.90 to 4.58]
  Week 68: number analyzed (Participants) | 10 | 33
  Week 68 | 0.68 [-3.81 to 5.17] | 1.25 [-1.32 to 3.83]
  Week 72: number analyzed (Participants) | 23 | 74
  Week 72 | -1.21 [-4.26 to 1.84] | 2.03 [0.14 to 3.92]
  Week 76: number analyzed (Participants) | 12 | 30
  Week 76 | 1.05 [-3.07 to 5.17] | 0.12 [-2.56 to 2.80]
  Week 80: number analyzed (Participants) | 23 | 75
  Week 80 | 0.47 [-2.58 to 3.52] | 2.32 [0.44 to 4.20]
  Week 84: number analyzed (Participants) | 8 | 30
  Week 84 | 3.21 [-1.77 to 8.19] | 1.56 [-1.12 to 4.25]
  Week 88: number analyzed (Participants) | 10 | 79
  Week 88 | 2.12 [-2.35 to 6.59] | 2.57 [0.72 to 4.42]
  Week 92: number analyzed (Participants) | 7 | 29
  Week 92 | -2.50 [-7.78 to 2.78] | 1.31 [-1.40 to 4.02]
  Week 96: number analyzed (Participants) | 16 | 63
  Week 96 | -0.03 [-3.61 to 3.55] | 2.96 [0.96 to 4.96]

17. Secondary Outcome: Change From Baseline in EORTC QLQ-C30 Global Health Status Score
Description: The EORTC-QLQ-C30 a 30-question tool was used to assess the overall QoL in cancer patients. It included 30 items resulting in 5 functional scales (physical, role, emotional, cognitive, and social functioning), 1 GHS scale, 3 symptom scales (fatigue, nausea and vomiting, and pain), and 6 single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). The questionnaire includes 28 items with 4-point Likert type responses from "1-not at all" to "4-very much" to assess functioning and symptoms; 2 items with 7-point Likert scales (1= poor and 7= excellent) for global health and overall QoL. Scores were transformed to a 0 to 100 scale, with higher scores representing better GHS, better functioning, and more symptoms.
Time Frame: as for outcome 15
Population: as for outcome 15
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on scale
Arm/Group | CyBorD | Daratumumab Plus CyBorD
Number analyzed (Participants) | 178 | 179
Score on scale
  Week 4: number analyzed (Participants) | 155 | 155
  Week 4 | -3.02 [-5.89 to -0.14] | -2.72 [-5.59 to 0.16]
  Week 8: number analyzed (Participants) | 146 | 152
  Week 8 | -4.15 [-7.09 to -1.21] | -3.83 [-6.73 to -0.93]
  Week 12: number analyzed (Participants) | 137 | 137
  Week 12 | -6.00 [-9.01 to -3.00] | -1.70 [-4.70 to 1.29]
  Week 16: number analyzed (Participants) | 130 | 132
  Week 16 | -7.17 [-10.23 to -4.11] | -2.75 [-5.78 to 0.28]
  Week 20: number analyzed (Participants) | 114 | 137
  Week 20 | -5.46 [-8.65 to -2.27] | -2.53 [-5.52 to 0.47]
  Week 24: number analyzed (Participants) | 33 | 127
  Week 24 | -4.26 [-9.43 to 0.92] | -0.76 [-3.83 to 2.31]
  Week 28: number analyzed (Participants) | 85 | 27
  Week 28 | -3.81 [-7.34 to -0.29] | -1.96 [-7.53 to 3.61]
  Week 32: number analyzed (Participants) | 15 | 105
  Week 32 | 3.03 [-4.33 to 10.39] | 1.36 [-1.90 to 4.62]
  Week 36: number analyzed (Participants) | 8 | 20
  Week 36 | 2.97 [-7.02 to 12.97] | 3.09 [-3.27 to 9.45]
  Week 40: number analyzed (Participants) | 12 | 100
  Week 40 | -6.13 [-14.31 to 2.05] | 5.10 [1.79 to 8.41]
  Week 44: number analyzed (Participants) | 9 | 19
  Week 44 | -1.37 [-10.79 to 8.05] | 0.16 [-6.36 to 6.68]
  Week 48: number analyzed (Participants) | 32 | 94
  Week 48 | -0.71 [-5.94 to 4.52] | 6.79 [3.40 to 10.17]
  Week 52: number analyzed (Participants) | 20 | 23
  Week 52 | -0.17 [-6.63 to 6.30] | 8.61 [2.64 to 14.59]
  Week 56: number analyzed (Participants) | 178 | 88
  Week 56 | 3.62 [-3.30 to 10.54] | 4.02 [0.56 to 7.49]
  Week 60: number analyzed (Participants) | 16 | 24
  Week 60 | 2.33 [-4.80 to 9.47] | 5.85 [-0.02 to 11.71]
  Week 64: number analyzed (Participants) | 12 | 81
  Week 64 | -5.49 [-13.67 to 2.70] | 8.27 [4.70 to 11.83]
  Week 68: number analyzed (Participants) | 10 | 34
  Week 68 | 6.19 [-2.75 to 15.14] | 4.95 [-0.08 to 9.99]
  Week 72: number analyzed (Participants) | 23 | 75
  Week 72 | -4.26 [-10.31 to 1.79] | 8.94 [5.27 to 12.60]
  Week 76: number analyzed (Participants) | 12 | 31
  Week 76 | 2.00 [-6.19 to 10.19] | 10.34 [5.11 to 15.57]
  Week 80: number analyzed (Participants) | 24 | 79
  Week 80 | 4.13 [-1.79 to 10.06] | 7.05 [3.45 to 10.65]
  Week 84: number analyzed (Participants) | 8 | 30
  Week 84 | 3.69 [-6.26 to 13.64] | 6.85 [1.54 to 12.15]
  Week 88: number analyzed (Participants) | 12 | 80
  Week 88 | -2.95 [-11.16 to 5.26] | 7.59 [4.01 to 11.16]
  Week 92: number analyzed (Participants) | 7 | 29
  Week 92 | 3.18 [-7.39 to 13.74] | 8.08 [2.70 to 13.45]
  Week 96: number analyzed (Participants) | 178 | 64
  Week 96 | 6.54 [-0.38 to 13.47] | 8.03 [4.15 to 11.91]

ADVERSE EVENTS:
Time Frame: All cause mortality: From baseline (Day -28) up to 7.1 years; Serious and Other AEs: For CyBorD: From start of treatment (Day 1) up to 30 days after last dose of study drug ( up to 8.33 months). Daratumumab plus CyBorD: From start of treatment (Day 1) up to 30 days after last dose of study drug ( up to 27.7 months).
Description: All cause mortality: All participants randomized into the study. Serious and Other AEs: Safety analysis set was defined as participants who have received at least 1 administration of any study treatment (partial or complete).
Arm/Group | Run-In: Daratumumab Plus CyBorD | CyBorD | Daratumumab Plus CyBorD
All-Cause Mortality (participants affected / at risk) | 11/28 | 67/193 | 47/195
Serious Adverse Events (participants affected / at risk) | 12/28 | 68/188 | 91/193
Other Adverse Events (participants affected / at risk) | 27/28 | 181/188 | 184/193
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Run-In: Daratumumab Plus CyBorD (N=28) | CyBorD (N=188) | Daratumumab Plus CyBorD (N=193)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Haemorrhagic Diathesis (Blood and lymphatic system disorders) | 0 | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Acute Left Ventricular Failure (Cardiac disorders) | 0 | 1 | 0
Acute Myocardial Infarction (Cardiac disorders) | 0 | 1 | 0
Angina Pectoris (Cardiac disorders) | 0 | 1 | 2
Arrhythmia (Cardiac disorders) | 0 | 2 | 0
Arteriospasm Coronary (Cardiac disorders) | 0 | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 0 | 2 | 6
Atrial Flutter (Cardiac disorders) | 0 | 0 | 2
Atrial Tachycardia (Cardiac disorders) | 0 | 1 | 0
Atrial Thrombosis (Cardiac disorders) | 0 | 1 | 0
Bradyarrhythmia (Cardiac disorders) | 0 | 0 | 1
Cardiac Arrest (Cardiac disorders) | 0 | 3 | 8
Cardiac Failure (Cardiac disorders) | 0 | 8 | 14
Cardiac Failure Congestive (Cardiac disorders) | 1 | 2 | 1
Cardiogenic Shock (Cardiac disorders) | 0 | 0 | 1
Cardiomyopathy (Cardiac disorders) | 0 | 1 | 0
Cardiovascular Insufficiency (Cardiac disorders) | 0 | 0 | 1
Coronary Artery Disease (Cardiac disorders) | 0 | 0 | 1
Left Ventricular Dysfunction (Cardiac disorders) | 0 | 0 | 1
Mitral Valve Incompetence (Cardiac disorders) | 0 | 1 | 0
Myocardial Infarction (Cardiac disorders) | 0 | 2 | 0
Pericarditis (Cardiac disorders) | 0 | 0 | 1
Sinus Bradycardia (Cardiac disorders) | 0 | 1 | 0
Sinus Node Dysfunction (Cardiac disorders) | 0 | 1 | 0
Sinus Tachycardia (Cardiac disorders) | 0 | 1 | 0
Supraventricular Tachycardia (Cardiac disorders) | 0 | 0 | 1
Hereditary Haemorrhagic Telangiectasia (Congenital, familial and genetic disorders) | 0 | 0 | 1
Amaurosis Fugax (Eye disorders) | 0 | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 0 | 1 | 1
Colitis Ischaemic (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 4 | 3
Gastric Haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Gastric Ulcer (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Intestinal Obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Melaena (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 2 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 3
Chest Pain (General disorders) | 0 | 1 | 0
Fatigue (General disorders) | 1 | 1 | 1
General Physical Health Deterioration (General disorders) | 0 | 1 | 0
Malaise (General disorders) | 0 | 1 | 1
Multiple Organ Dysfunction Syndrome (General disorders) | 1 | 0 | 0
Non-Cardiac Chest Pain (General disorders) | 0 | 1 | 1
Oedema (General disorders) | 1 | 0 | 0
Oedema Peripheral (General disorders) | 1 | 2 | 3
Peripheral Swelling (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 1
Sudden Cardiac Death (General disorders) | 0 | 1 | 1
Sudden Death (General disorders) | 0 | 3 | 6
Bile Duct Stone (Hepatobiliary disorders) | 0 | 0 | 1
Hepatomegaly (Hepatobiliary disorders) | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 1
Adenovirus Infection (Infections and infestations) | 0 | 0 | 1
Biliary Sepsis (Infections and infestations) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1 | 0
Candida Sepsis (Infections and infestations) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 2 | 1 | 2
Escherichia Bacteraemia (Infections and infestations) | 0 | 0 | 1
Gastrointestinal Infection (Infections and infestations) | 0 | 1 | 0
Herpes Zoster (Infections and infestations) | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 2 | 1
Lower Respiratory Tract Infection (Infections and infestations) | 0 | 3 | 1
Lower Respiratory Tract Infection Viral (Infections and infestations) | 0 | 0 | 1
Neutropenic Sepsis (Infections and infestations) | 0 | 0 | 1
Orchitis (Infections and infestations) | 0 | 0 | 1
Peritonitis (Infections and infestations) | 1 | 0 | 1
Pneumonia (Infections and infestations) | 2 | 9 | 14
Pneumonia Pneumococcal (Infections and infestations) | 0 | 1 | 1
Pulmonary Sepsis (Infections and infestations) | 0 | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 0 | 1
Pyelonephritis Acute (Infections and infestations) | 0 | 0 | 1
Respiratory Syncytial Virus Infection (Infections and infestations) | 0 | 0 | 1
Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 1
Respiratory Tract Infection Viral (Infections and infestations) | 0 | 0 | 1
Rhinovirus Infection (Infections and infestations) | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 7
Septic Shock (Infections and infestations) | 0 | 1 | 2
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 1 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 4
Wound Infection (Infections and infestations) | 0 | 0 | 1
Delayed Engraftment (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 3 | 0 | 0
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Head Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Hip Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Rib Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Skin Laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0
Traumatic Liver Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Influenza A Virus Test Positive (Investigations) | 0 | 0 | 1
Weight Decreased (Investigations) | 0 | 0 | 1
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 2 | 2
Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1
Failure to Thrive (Metabolism and nutrition disorders) | 0 | 0 | 1
Fluid Overload (Metabolism and nutrition disorders) | 0 | 5 | 1
Hyperglycaemic Hyperosmolar Nonketotic Syndrome (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 3 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Connective Tissue Inflammation (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Myopathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Cerebrovascular Accident (Nervous system disorders) | 0 | 1 | 1
Facial Paralysis (Nervous system disorders) | 0 | 0 | 1
Hemiparesis (Nervous system disorders) | 0 | 0 | 1
Ischaemic Stroke (Nervous system disorders) | 0 | 1 | 0
Peripheral Sensorimotor Neuropathy (Nervous system disorders) | 0 | 0 | 1
Status Epilepticus (Nervous system disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 1 | 6 | 4
Anxiety (Psychiatric disorders) | 0 | 2 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 1
Depressed Mood (Psychiatric disorders) | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 1 | 0
Mental Status Changes (Psychiatric disorders) | 1 | 0 | 0
Suicide Attempt (Psychiatric disorders) | 1 | 0 | 0
Acute Kidney Injury (Renal and urinary disorders) | 3 | 1 | 3
Chronic Kidney Disease (Renal and urinary disorders) | 0 | 1 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0
Nephropathy (Renal and urinary disorders) | 0 | 0 | 1
Nephrotic Syndrome (Renal and urinary disorders) | 0 | 0 | 1
Renal Failure (Renal and urinary disorders) | 0 | 2 | 1
Renal Impairment (Renal and urinary disorders) | 0 | 1 | 0
Female Genital Tract Fistula (Reproductive system and breast disorders) | 0 | 0 | 1
Acute Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Lung Disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 4
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pulmonary Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin Mass (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Elective Surgery (Surgical and medical procedures) | 0 | 0 | 1
Circulatory Collapse (Vascular disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 1 | 1
Orthostatic Hypotension (Vascular disorders) | 0 | 0 | 1
Thrombosis (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Run-In: Daratumumab Plus CyBorD (N=28) | CyBorD (N=188) | Daratumumab Plus CyBorD (N=193)
Anaemia (Blood and lymphatic system disorders) | 13 | 44 | 49
Eosinopenia (Blood and lymphatic system disorders) | 2 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 2 | 1 | 1
Leukopenia (Blood and lymphatic system disorders) | 5 | 7 | 11
Lymphopenia (Blood and lymphatic system disorders) | 12 | 28 | 37
Neutropenia (Blood and lymphatic system disorders) | 3 | 12 | 21
Thrombocytopenia (Blood and lymphatic system disorders) | 7 | 21 | 34
Palpitations (Cardiac disorders) | 1 | 6 | 12
Tinnitus (Ear and labyrinth disorders) | 2 | 0 | 4
Dry Eye (Eye disorders) | 4 | 2 | 5
Ocular Hyperaemia (Eye disorders) | 2 | 2 | 2
Vision Blurred (Eye disorders) | 5 | 8 | 13
Abdominal Distension (Gastrointestinal disorders) | 3 | 12 | 15
Abdominal Pain (Gastrointestinal disorders) | 5 | 17 | 21
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 13 | 18
Ascites (Gastrointestinal disorders) | 2 | 2 | 4
Constipation (Gastrointestinal disorders) | 12 | 54 | 70
Diarrhoea (Gastrointestinal disorders) | 19 | 55 | 69
Dry Mouth (Gastrointestinal disorders) | 2 | 6 | 5
Dyspepsia (Gastrointestinal disorders) | 1 | 12 | 8
Flatulence (Gastrointestinal disorders) | 2 | 0 | 7
Gastrointestinal Pain (Gastrointestinal disorders) | 2 | 1 | 0
Nausea (Gastrointestinal disorders) | 12 | 51 | 55
Stomatitis (Gastrointestinal disorders) | 3 | 5 | 4
Vomiting (Gastrointestinal disorders) | 5 | 21 | 29
Asthenia (General disorders) | 2 | 20 | 31
Chills (General disorders) | 1 | 4 | 10
Fatigue (General disorders) | 16 | 52 | 55
Injection Site Bruising (General disorders) | 2 | 0 | 4
Injection Site Discolouration (General disorders) | 2 | 1 | 2
Injection Site Erythema (General disorders) | 5 | 21 | 18
Non-Cardiac Chest Pain (General disorders) | 2 | 8 | 3
Oedema Peripheral (General disorders) | 14 | 66 | 71
Pyrexia (General disorders) | 3 | 15 | 26
Hyperbilirubinaemia (Hepatobiliary disorders) | 5 | 9 | 4
Bronchitis (Infections and infestations) | 4 | 5 | 11
Cellulitis (Infections and infestations) | 2 | 4 | 3
Conjunctivitis (Infections and infestations) | 1 | 5 | 12
Herpes Zoster (Infections and infestations) | 0 | 12 | 13
Hordeolum (Infections and infestations) | 0 | 11 | 9
Nasopharyngitis (Infections and infestations) | 0 | 11 | 20
Pneumonia (Infections and infestations) | 1 | 6 | 13
Rhinitis (Infections and infestations) | 1 | 2 | 10
Sinusitis (Infections and infestations) | 3 | 2 | 6
Tooth Infection (Infections and infestations) | 2 | 1 | 4
Upper Respiratory Tract Infection (Infections and infestations) | 10 | 21 | 50
Urinary Tract Infection (Infections and infestations) | 1 | 6 | 14
Contusion (Injury, poisoning and procedural complications) | 6 | 6 | 15
Fall (Injury, poisoning and procedural complications) | 4 | 8 | 15
Skin Laceration (Injury, poisoning and procedural complications) | 3 | 3 | 4
Alanine Aminotransferase Increased (Investigations) | 6 | 10 | 21
Aspartate Aminotransferase Increased (Investigations) | 7 | 8 | 20
Basophil Count Increased (Investigations) | 2 | 0 | 0
Blood Alkaline Phosphatase Increased (Investigations) | 5 | 11 | 10
Blood Creatinine Increased (Investigations) | 7 | 16 | 20
Gamma-Glutamyltransferase Increased (Investigations) | 0 | 11 | 13
Hepatic Enzyme Increased (Investigations) | 2 | 0 | 0
Monocyte Count Increased (Investigations) | 3 | 0 | 0
Weight Decreased (Investigations) | 1 | 6 | 11
Weight Increased (Investigations) | 4 | 6 | 9
Decreased Appetite (Metabolism and nutrition disorders) | 5 | 22 | 21
Hypercalcaemia (Metabolism and nutrition disorders) | 3 | 2 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 10 | 7 | 12
Hyperkalaemia (Metabolism and nutrition disorders) | 3 | 7 | 14
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 8 | 14
Hypoalbuminaemia (Metabolism and nutrition disorders) | 7 | 11 | 9
Hypocalcaemia (Metabolism and nutrition disorders) | 6 | 9 | 13
Hypoglycaemia (Metabolism and nutrition disorders) | 6 | 3 | 7
Hypokalaemia (Metabolism and nutrition disorders) | 7 | 28 | 26
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 | 3 | 6
Hyponatraemia (Metabolism and nutrition disorders) | 7 | 6 | 16
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 9 | 23
Back Pain (Musculoskeletal and connective tissue disorders) | 3 | 11 | 28
Joint Swelling (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 10 | 19
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 5 | 11 | 16
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 7 | 17
Neck Pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 3
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 5 | 9 | 24
Dizziness (Nervous system disorders) | 13 | 26 | 31
Dysgeusia (Nervous system disorders) | 6 | 11 | 15
Headache (Nervous system disorders) | 6 | 18 | 30
Hypoaesthesia (Nervous system disorders) | 5 | 3 | 7
Memory Impairment (Nervous system disorders) | 2 | 2 | 1
Neuralgia (Nervous system disorders) | 0 | 5 | 10
Paraesthesia (Nervous system disorders) | 5 | 12 | 17
Peripheral Sensory Neuropathy (Nervous system disorders) | 5 | 37 | 65
Syncope (Nervous system disorders) | 1 | 9 | 14
Tremor (Nervous system disorders) | 0 | 2 | 12
Anxiety (Psychiatric disorders) | 0 | 11 | 12
Confusional State (Psychiatric disorders) | 3 | 1 | 2
Depression (Psychiatric disorders) | 3 | 6 | 9
Insomnia (Psychiatric disorders) | 9 | 47 | 49
Haematuria (Renal and urinary disorders) | 2 | 0 | 6
Pollakiuria (Renal and urinary disorders) | 5 | 4 | 3
Renal Impairment (Renal and urinary disorders) | 2 | 11 | 10
Urinary Incontinence (Renal and urinary disorders) | 2 | 0 | 1
Urinary Retention (Renal and urinary disorders) | 2 | 0 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 19 | 35
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 | 29 | 46
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 4 | 6 | 8
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 10
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 12
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 5 | 5 | 15
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 13
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 2
Dry Skin (Skin and subcutaneous tissue disorders) | 5 | 2 | 12
Erythema (Skin and subcutaneous tissue disorders) | 4 | 3 | 12
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 8 | 16
Rash (Skin and subcutaneous tissue disorders) | 4 | 13 | 19
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 5 | 2 | 8
Rash Pruritic (Skin and subcutaneous tissue disorders) | 2 | 1 | 2
Flushing (Vascular disorders) | 2 | 3 | 2
Hot Flush (Vascular disorders) | 2 | 1 | 3
Hypertension (Vascular disorders) | 2 | 3 | 14
Hypotension (Vascular disorders) | 6 | 21 | 30
Orthostatic Hypotension (Vascular disorders) | 1 | 11 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2019-10-10): https://cdn.clinicaltrials.gov/large-docs/65/NCT03201965/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-04): https://cdn.clinicaltrials.gov/large-docs/65/NCT03201965/SAP_001.pdf